CLINICAL TRIAL: NCT05535855
Title: Phase 1/1b Safety and Tolerability Trial of CD19 Directed CAR T Cells in Adult Patients With B-Cell Acute Lymphoblastic Leukemia (B-ALL) With Minimal Residual Disease (MRD) Positivity at First Complete Remission
Brief Title: UCD19 CAR T Therapy in Adults With B-ALL and MRD Positivity in CR1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-0054.cc; NCI-2023-05480 (Other: CTRP)
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoid Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UCD19 CAR T Infusion (Experimental): Lymphodepleting chemotherapy followed by infusion of UCD19 CAR T cells. Infusion is subject to a seven (7) day delay following chemotherapy completion if needed for resolution of clinical toxicities or to allow for product release.
  Interventions: Drug: CD19 Directed CAR T Cell

INTERVENTIONS:
Drug: CD19 Directed CAR T Cell — The UCD19 CAR T cells are developed through transfection of autologous peripheral blood mononuclear cells with a lentivirus carrying the DNA that encodes a short chain fragment variable region (scFv) derived from an anti-CD19 monoclonal antibody, among other elements.
  Other Names: UCD19 CAR T cells

SUMMARY:
This open-label, single arm Phase 1/1b trial aims to determine the safety and tolerability of anti-CD19 chimeric antigen receptor-expressing (CAR) T cells (UCD19 CAR T) in adults with B-ALL that are in first complete remission with MRD positivity. This trial will enroll 10 patients during Phase 1 for apheresis, treatment with lymphodepleting chemotherapy, and UCD19 CAR T cell infusion. Patients will be assessed for DLTs (within 42 days after CAR T infusion) to determine a maximum tolerated dose (MTD), duration of B cell aplasia, overall response rate (at 1-3-, 6- and 12-months), and overall survival and event free survival (at 12- and 24- months) post UCD19 CAR T infusion.

After the initial dose escalation phase, an additional 12 participants will be enrolled in the dose expansion at the MTD to determine preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years of age with no upper age limit
2. ECOG Performance Status ≤ 2
3. Confirmed B-cell ALL in first complete morphologic remission
4. MRD positivity as defined by:

   1. For Ph- ALL: > 0.01% by FACS or > 0 clonal sequences by NGS (clonoSEQ). MRD assessment for eligibility must be at least 28 days after the start of SOC induction therapy. Remission-induction therapy must have consisted of multi-agent chemotherapy (≥ 3 systemic anti-leukemia chemotherapy agents).
   2. For Ph+ ALL: > 0.01% by FACS, > 0 clonal sequences by NGS (clonoSEQ), or less than complete molecular remission (undetectable BCR-ABL1 transcripts by RT-PCR assay with sensitivity of at least 1 in 100,000). MRD assessment for eligibility must be at least 57 days after the start of SOC induction therapy. Remission-induction therapy must have consisted of a BCR-ABL1 directed tyrosine kinase inhibitor and at least one other systemic anti-leukemia chemotherapy agent.
5. Peripheral blood CD3 count must be > 0.15 x 106 cells/mL within 21 days prior to proceeding with apheresis.
6. Toxicities from prior therapy must be stable and recovered to ≤ Grade 2 (exceptions include non-clinically significant toxicities such as alopecia and the organ function definitions provided in inclusion criteria 7).
7. Adequate organ function as defined by:

   1. Absolute neutrophil count (ANC) ≥ 500/μL.
   2. Platelet count ≥ 50,000/μL.
   3. Renal: Either Creatinine ≤ 2 mg/dL OR creatinine clearance (as estimated by Cockcroft Gault equation) ≥ 60 mL/min.
   4. Hepatic: Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 2.5 upper limit of normal (ULN).
   5. Total bilirubin ≤ 1.5 mg/dL, except in subjects with Gilbert's syndrome where a bilirubin < 3.0 mg/dL will be acceptable.
   6. Cardiac: Ejection fraction ≥ 45%, no evidence of physiologically significant pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings at the time of screening.
   7. Pulmonary: No clinically significant pleural effusion.

   i. Baseline oxygen saturation > 92% on room air and; ii. Pulmonary Function Test: Diffuse capacity of the lungs for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) are all ≥50% of predicted by spirometry after correcting for hemoglobin.
8. Females of childbearing potential must have a negative serum pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
9. Subjects of childbearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for 12 months after receiving the UCD19 infusion.
10. Must be able to give informed consent; subjects unable to give informed consent will not be eligible for this study.
11. Be able to consent to long-term follow-up protocol (#20-0188).

Exclusion Criteria:

1. Previous CAR T therapy.
2. Relapsed or refractory B-cell acute lymphoblastic leukemia, including patients who have evidence of MRD after having previously documented MRD-negative remission.
3. Mixed phenotype acute leukemia or Burkitt's lymphoma
4. Not in hematological remission at time of enrollment (Remission is defined as < 5% blasts)
5. Signs or symptoms of active CNS disease or detectable evidence of CNS disease on MRI at the time of screening. Subjects who have been previously treated for CNS disease but have no evidence of disease at screening are eligible.
6. History of malignancy unless disease free for at least 3 years. Exceptions include non-melanoma skin cancer or carcinoma in situ (e.g., cervix, bladder, breast).
7. Uncontrolled fungal, bacterial, viral, or other infection requiring antimicrobials for management; simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
8. Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (hepatitis B surface antigen [HBsAg] positive) or hepatitis C.
9. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment or have cardiac atrial or cardiac ventricular lymphoma involvement.
10. Venous thrombosis or embolism not managed on a stable regimen of anticoagulation.
11. Any medical condition that in the judgement of the Sponsor is likely to interfere with assessment of safety or efficacy of study treatment.
12. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
13. Females planning to become pregnant during the course of the study.

Apheresis Eligibility In order to proceed with apheresis, enrolled participants must continue to meet all inclusion criteria within no more than 21 days prior to apheresis, unless otherwise specified.

Note: Disease evaluation to meet inclusion criteria must be completed within 30 days prior to apheresis.

Screening Eligibility In order to proceed, participants must meet all inclusion criteria. Medical history, blood tests, and assessments may be done as standard of care but must be performed within 14 to 30 days prior to enrollment unless otherwise indicated.

Lymphodepleting Chemotherapy Eligibility

In order to proceed with lymphodepleting chemotherapy, enrolled participants must have all assessments below completed, and continue to meet all inclusion criteria within 72 hours of initiation of lymphodepletion, with the following clarifications:

* Disease restaging studies will be performed as clinically indicated but must be within 14 days prior to initiation of lymphodepletion.
* Peripheral blood for CD3 count must be obtained within 21 days prior to apheresis and, therefore, is not applicable for determining lymphodepleting chemotherapy eligibility.
* In lieu of exclusion criteria #4, there must be no evidence of rapidly progressive disease prior to LD chemotherapy initiation per Investigator assessment.

Bridging disease directed antineoplastic therapy is allowed with progressive disease after enrollment but before initiation of lymphodepleting chemotherapy will be removed from the study.

The following assessments will be used to confirm that the participant is able to initiate lymphodepleting chemotherapy (within 72 hours of starting chemotherapy):

* Medical history and Baseline Abnormalities

  * Medical history (defined as ongoing medical conditions identified before the subject's first study-specific intervention (i.e., initiation of LD Chemotherapy on Day -5).
  * Baseline abnormalities refer to abnormal clinical findings (e.g., laboratory values, vital signs, ECG results, etc.) identified before the start of LD Chemotherapy that may or may not be related to the subject's underlying disease.
  * All medical history and baseline abnormalities should be entered in the eCRF. Events should be assessed within 30 days prior to enrollment until LD Chemotherapy. Grading per CTCAE v5.0 should reflect the patient's status at the time of LD Chemotherapy.
* Physical exam

UCD19 CAR T Cell Infusion Eligibility

Participants must meet the following criteria in order for cells to be infused (based on labs obtained within 24 hours of cell infusion):

* UCD19 CAR T Cells must have met release criteria.
* Performance status determination (ECOG must be ≤ 2).
* Participant remains clinically stable without evidence of vital sign instability.
* Must not have ALT/SGPT and AST/SGOT > 10x the ULN or bilirubin >2x the ULN, (unless history of Gilberts syndrome where bilirubin must not be >3x ULN).
* Adequate renal function as defined in the Inclusion Criteria.
* No evidence of uncontrolled infection within 48 hours prior to cell infusion as determined by the PI or sub-investigator. If these criteria are not met, measures will be taken to resolve the underlying condition(s). If successful, cells may be infused up to (and including) 7 days following the time of the planned infusion with no additional lymphodepletion. If the UCD19 CAR T Cell infusion is delayed greater than 7 days, lymphodepleting chemotherapy MAY be repeated. Prior to commencing a second round of lymphodepletion, participants must meet lymphodepletion criteria described above.

Prior to moving to the treatment portion of this study, participants must meet limited eligibility criteria as specified above.

UCD19 CAR T cells may be infused on an inpatient or outpatient basis at the discretion of the treating investigator. Following discharge, participants will continue with once-a-week evaluation until Day 42. If UCD19 CAR T cells are infused on an outpatient basis or following discharge after being inpatient, the participant will need to stay within 1 hour of the Anschutz Medical Campus for at least 4 weeks from date of CAR T cell infusion for monitoring by the treating investigator.

TKI Therapy Post ICD19 CAR T Cell Infusion Eligibility

Participants must meet the following criteria in order to receive TKI therapy:

* Disease classified as Ph+ B-ALL.
* Must be past the DLT period (Day 42).
* Platelet count > 50,000/μL.
* ANC > 1000/μL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of UCD19 CAR T in Adults With B-ALL in first complete remission with MRD Positivity: occurrence and frequency of Adverse Events (AEs) | Up to 30 days after last day of study participation
  The occurrence and frequency of Adverse Events will be graded using the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grading criteria.
Safety of UCD19 CAR T in Adults With B-ALL in first complete remission with MRD Positivity: occurrence of Dose Limiting Toxicities (DLTs) | 42 days
  Adverse events that are at least possibly related to the UCD19 CAR T cells with onset within the first 42 days following UCD19 CAR T cell infusion and are ≥ Grade 3 in severity will be considered DLTs.
  With exception to hematological toxicity for subjects with normal, Grade 1 or Grade 2 Hematologic Parameters at baseline (independent of transfusion) and cytopenias NOT due to Bone Marrow Involvement by Disease. However, any Grade 4 hematological toxicity (i.e., neutropenia or thrombocytopenia with the exception of lymphopenia) persisting beyond 42 days after infusion will be considered a DLT unless toxicity is attributed to patient's underlying disease.
Preliminary efficacy of UCD19 CAR T infusion at the MTD in adult B-ALL patients at first complete remission with MRD positivity | 12 and 24 months
  Determine the Relapse Free Survival (RFS) rate post UCD19 CAR T infusion. RFS will be measured from the date of infusion of the UCD19 CAR T product to the time of relapse or death from any cause

SECONDARY OUTCOMES:
Overall response rate (ORR) at 1, 3, 6, 12, and 24 months post UCD19 CAR T infusion as measured by MRD. | 1, 3, 6, 12, and 24 months
  MRD negativity is defined as bone marrow that has no detectable blasts at or above the sensitivity threshold for the particular assay used (approximately 0.01% for FACS-MRD, 0.001% for BCR-ABL qPCR, 0.0001% for IgH/TCR NGS).
  MRD positivity post UCD19 CAR T infusion is defined as > 0.01% by FACS or a rising number of > 0 clonal sequences by NGS (clonoSEQ) at two timepoints at least 2-4 weeks apart in the bone marrow or peripheral blood for Ph- ALL, and either > 0.01% by FACS, a rising number of > 0 clonal sequences by NGS (clonoSEQ), or less than complete molecular remission (undetectable BCR-ABL1 transcripts by quantitative PCR assay with sensitivity of at least 1 in 100,000) at two timepoints at least 2-4 weeks apart in the bone marrow or peripheral blood for Ph+ ALL.
Overall Survival (OS) at 12 and 24 months post UCD19 CAR T infusion. | 12 and 24 months
  OS defined as measured from the date of infusion to the time of death from any cause.
Event Free Survival (EFS) at 12 and 24 months post UCD19 CAR T infusion | 12 and 24 months
  EFS is defined as failure to achieve MRD-negativity (approximately 0.01% for FACS-MRD, 0.001% for BCR-ABL qPCR), disease relapse, or death from any cause from the date of infusion

OTHER OUTCOMES:
Duration of B-cell aplasia | 12 months
  B-cell aplasia defined as <3.0% CD19+ cells/total lymphocytes by peripheral blood flow cytometry.
Assessment of minimal residual disease by next generation sequencing | 1, 3, 6, and 12 months
  MRD by next generation sequencing for clonal B-cell receptor gene rearrangements

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schwartz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No